CLINICAL TRIAL: NCT00228436
Title: A Phase 2, Open-label, Multi-center, Sequential Dose Finding Study of the Safety, Pharmacodynamics, and Pharmacokinetics of Multiple Doses of Subcutaneously Administered Peginesatide in Chronic Kidney Disease Patients Not on Dialysis and Not on Erythropoiesis Stimulating Agent (ESA) Treatment
Brief Title: Safety, PD & PK of Multiple Doses of Peginesatide for Anemia in Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-04; 2005-002218-39 (EudraCT Number)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (Experimental): Peginesatide starting dose of 0.05 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 6 doses.
  Interventions: Drug: peginesatide
- Cohort 2 (Experimental): Peginesatide starting dose of 0.075 mg/kg administered SC Q4W for a total of 6 doses.
  Interventions: Drug: peginesatide
- Cohort 3 (Experimental): Peginesatide starting dose of 0.025 mg/kg administered SC Q4W for a total of 6 doses.
  Interventions: Drug: peginesatide
- Cohort 4 (Experimental): Peginesatide starting dose of 0.05 mg/kg administered intravenously (IV) Q4W for a total of 6 doses.
  Interventions: Drug: peginesatide
- Cohort 5 (Experimental): Peginesatide starting dose of 0.025 mg/kg administered SC once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Drug: peginesatide
- Cohort 6 (Experimental): Peginesatide starting dose of 0.0375 mg/kg administered SC Q2W for a total of 12 doses.
  Interventions: Drug: peginesatide
- Cohort 7 (Experimental): Peginesatide fixed starting dose of 4 mg administered SC Q4W for a total of 6 doses.
  Interventions: Drug: peginesatide
- Cohort 8 (Experimental): Peginesatide fixed starting dose of 3 mg administered SC Q4W for a total of 6 doses.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide
  Other Names: Omontys; Hematide; AF37702 Injection

SUMMARY:
The purpose of this study was to evaluate the safety, pharmacodynamics (PD), and pharmacokinetics (PK) of multiple subcutaneous injections of peginesatide in participants with chronic kidney disease (CKD) not on dialysis who had not received erythropoiesis stimulating agent (ESA) treatment.

DETAILED DESCRIPTION:
This was a Phase 2, dose finding study designed to evaluate peginesatide treatment of participants with CKD not on ESA treatment. The objective was to determine the range of doses of peginesatide administered subcutaneously once every 4 weeks (Q4W) that increased and maintained hemoglobin at 11 to 13 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local and national guidelines;
* Males or females ≥ 18 and ≤ 85 years of age. Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice an adequate form of contraception for at least 4 weeks prior to study start, and must be willing to continue contraception for at least 4 weeks after the last dose of study drug;
* Chronic kidney disease stage 3 or 4 (estimated Glomerular filtration rate [GFR] of 15-60 mL/min within 28 days prior to study drug administration) and not expected to begin dialysis for at least 12 weeks;
* Two hemoglobin values of ≥ 9.0 and < 11.0 g/dL within 14 days prior to study drug administration, including at least one of the values drawn within 7 days prior to study drug administration;
* One serum ferritin level ≥ 100 micrograms per liter (μg/L) and transferrin saturation ≥ 20 % within 4 weeks prior to study drug administration;
* One serum or red cell folate level above lower limit of normal within 4 weeks prior to study drug administration;
* One vitamin B12 level above lower limit of normal within 4 weeks prior to study drug administration;
* Weight ≥ 45 kg within 4 weeks prior to study drug administration;
* One white blood cell count ≥ 3.0 x 10^9/L within 4 weeks prior to study drug administration; and
* One platelet count ≥ 100 x 10^9/L within 4 weeks prior to study drug administration.

Exclusion Criteria:

* Prior treatment with any erythropoiesis stimulating agent in the 12 weeks prior to study drug administration;
* Any prior treatment with Eprex®;
* Known intolerance to any erythropoiesis stimulating agent;
* History of antibodies to any erythropoiesis stimulating agent or history of pure red cell aplasia;
* Prior hemodialysis or peritoneal dialysis treatment;
* Known intolerance to parenteral iron supplementation;
* Red blood cell transfusion within 12 weeks prior to study drug administration;
* Hemoglobinopathy [e.g., homozygous sickle-cell disease (sickle-cell trait does not exclude patient), thalassemia of all types, etc.];
* Known hemolysis;
* Chronic, uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.);
* C Reactive Protein (CRP) greater than 30 mg/L within the 4 weeks prior to study drug administration;
* Febrile illness within 7 days prior to study drug administration;
* Uncontrolled or symptomatic secondary hyperparathyroidism;
* Poorly controlled hypertension within 4 weeks prior to study drug administration, per Investigator's clinical judgment (e.g. systolic ≥ 170mm Hg, diastolic ≥ 100 mm Hg on repeat readings);
* Epileptic seizure in the 6 months prior to study drug administration;
* Chronic congestive heart failure (New York Heart Association Class IV);
* High likelihood of early withdrawal or interruption of the study;
* Evidence of malignancy within the past 5 years (except non-melanoma skin cancer which is not an exclusion criterion);
* Life expectancy < 12 months;
* Anticipated elective surgery during the study period; and
* Previous exposure to any investigational agent within 6 weeks prior to administration of study drug or planned receipt during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who achieved a target hemoglobin response during the study. | 25 weeks
  A target hemoglobin response is defined as a hemoglobin increase of ≥ 1.0 gram per deciliter (g/dL) from baseline and a hemoglobin value ≥ 11.0 g/dL during the study.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | 25 weeks
Pharmacokinetic parameters | 25 weeks
Percentage of participants with hemoglobin values in the range of 11.0 to 13.0 g/dL throughout the study. | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Affymax, Study Director — Affymax, Inc
Locations (13):
- Poland (6):
  - Research Facility, Bialystok
  - Research Facility, Gdansk
  - Research Facility, Katowice
  - Research Facilities, Krakow
  - Research Facility, Lodz
  - Research Facility, Warsaw
- United Kingdom (7):
  - Research Facility, Coventry
  - Research Facility, Croydon
  - Research Facility, Derby
  - Research Facility, Leicester
  - Research Facilities, London
  - Research Facility, Salford
  - Research Facility, Swansea

REFERENCES:
- [Derived] Macdougall IC, Wiecek A, Tucker B, Yaqoob M, Mikhail A, Nowicki M, MacPhee I, Mysliwiec M, Smolenski O, Sulowicz W, Mayo M, Francisco C, Polu KR, Schatz PJ, Duliege AM. Dose-finding study of peginesatide for anemia correction in chronic kidney disease patients. Clin J Am Soc Nephrol. 2011 Nov;6(11):2579-86. doi: 10.2215/CJN.10831210. Epub 2011 Sep 22. PMID 21940838